CLINICAL TRIAL: NCT05656625
Title: Comparison of Ultrasound-guided Brachial Plexus Blocks and Selective Distal Blocks in Terms of Anesthesia Success and Discharge Time in Hand and Wrist Surgeries: A Single Center, Historic Cohort Study
Brief Title: Comparison of Ultrasound-guided Brachial Plexus Blocks and Selective Distal Blocks in Terms of Anesthesia
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Gamze Ertas, principle investigator, Samsun University
Other Study IDs: distal block
Record Dates: First submitted 2022-11-21; First posted 2022-12-19 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Pain, Postoperative; Anesthesia, Local; Patient Satisfaction
Keywords: distal nerve block,patient satisfaction,hand surgery
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group distal nerve block(DNB): Radial, median and ulnar nerve blocks were used alone or in combinations as a method of anesthesia for patients who had undergone hand and wrist surgery.
  Interventions: Other: descriptive
- group brachial plexus block(BPB): Brachial plexus blocks (infraclavicular, axillary etc.) was applied to patients who were going to undergo hand and wrist surgery.
  Interventions: Other: descriptive

INTERVENTIONS:
Other: descriptive — The block performed (distal peripheral nerve block and/or brachial nerve block) and the volume applied, block performance time, first analgesia times, surgery times, surgery types, discharge times, presence of additional complaints will be recorded. The data obtained by grouping the patients according to the type of anesthesia applied (brachial plexus block and distal nerve blocks) will be subjected to statistical analysis.

SUMMARY:
Ultrasound-guided brachial plexus blocks (infraclavicular, axillary) can be applied as the main anesthetic method in hand and wrist surgeries, as well as single or combination block applications of the median, radial and ulnar nerves at the forearm level.

Here, we aimed to retrospectively evaluate the perioperative and postoperative data of patients who underwent hand and wrist surgery under distal nerve blocks and brachial plexus blocks in our hospital.

DETAILED DESCRIPTION:
The retrospective files of patients who used ultrasound guided regional anesthesia techniques as the main anesthetic method in hand and wrist surgeries in our hospital between 01.01.2021 and 01.09.2022 will be examined. Patients over the age of 18 who go to hand and wrist surgery will be included. Patients who have undergone surgical intervention in more than one region in the same session and who have psychiatric disorders that will affect the perception of pain will be excluded from the study. Demographic characteristics, American Society of Anesthesiology (ASA) scores, comorbidity, block performed (distal peripheral nerve block and/or brachial nerve block) and volume applied, block performance time, first analgesia times, surgery times, surgery types, discharge times, additional The existence of the complaint will be recorded. The data obtained by grouping the patients according to the type of anesthesia applied (brachial plexus block and distal nerve blocks) will be subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who go to hand and wrist surgery will be included.

Exclusion Criteria:

* Patients who have undergone surgical intervention in more than one region in the same session and who have psychiatric disorders that will affect the perception of pain will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who go to hand and wrist surgery will be included.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Quality in Anaesthesia | up 24 hours
  The patients were called by phone and asked to evaluate the anesthesia technique used in their surgery. Three main judgments including 'quality of anesthesia', 'whether they would prefer the same anesthesia again' and 'whether they would recommend this technique to others' were evaluated with a 5-point Likert scale. 5 point Likert scale consists of 5 answer options which will contain two extreme poles and a neutral option connected with intermediate answer options. In evaluation of parient satisfaction, we used 5 point Likert scale example to measure satisfaction is:
  (1) Very dissatisfied, (2)Dissatisfied, (3) Neither satisfied nor dissatisfied, (4) Satisfied , (5)Very satisfied .
  In other terms, (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.

SECONDARY OUTCOMES:
discharge time | up to 24 hours
  The time of discharge will be specified in both groups.
block performance time | intraoperative
  Block performance time was defined as the time from ultrasound probe insertion to needle removal at the end of perineural injections.
additional anesthetic/analgesic requirement | perioperative period
  additional analgesic requirement will be evaluated intraoperatively or postoperatively.
complications | up to 24 hours
  The presence of complications will be evaluated during and after the block.

CONTACTS AND LOCATIONS:
Overall Officials: gamze MD ertaş, specialist, Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Ilkadım, Turkey (Türkiye)

REFERENCES:
- [Result] Soberon JR Jr, Crookshank JW 3rd, Nossaman BD, Elliott CE, Sisco-Wise LE, Duncan SF. Distal Peripheral Nerve Blocks in the Forearm as an Alternative to Proximal Brachial Plexus Blockade in Patients Undergoing Hand Surgery: A Prospective and Randomized Pilot Study. J Hand Surg Am. 2016 Oct;41(10):969-977. doi: 10.1016/j.jhsa.2016.07.092. Epub 2016 Aug 11. PMID 27524691
- [Result] Ince I, Aksoy M, Celik M. Can We Perform Distal Nerve Block Instead of Brachial Plexus Nerve Block Under Ultrasound Guidance for Hand Surgery? Eurasian J Med. 2016 Oct;48(3):167-171. doi: 10.5152/eurasianjmed.2016.0256. PMID 28149139